CLINICAL TRIAL: NCT02156206
Title: Building Capacity of State and Local Actors to Respond to Violence Against Women: Impact Evaluation of the 123 Women Emergency Phone Line in Medellín (Colombia), Component of the Program "Seguridad Pública".
Brief Title: Impact Evaluation of the 123 Women Emergency Phone Line in Medellín, Colombia
Status: Completed | Type: Observational
Sponsor: Econometría Consultores (Other)
Collaborators: Inter-American Development Bank (Other)
Responsible Party: Sponsor
Other Study IDs: ATN/MG-13064-RG ECO 577-2
Record Dates: First submitted 2014-06-03; First posted 2014-06-05 (Estimated); Last update posted 2017-02-07 (Estimated); Status verified 2017-02

CONDITIONS: Violence Against Women (VAW)

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (2):
- 123 women line: Women who call the 123 emergency line and have also immediate services from the 123 women emergency line
  Interventions: Behavioral: 123 women emergency phone line in Medellin, Colombia
- No treatment: Women who call the 123 emergency line and do not have immediate services from the 123 women emergency line

INTERVENTIONS:
Behavioral: 123 women emergency phone line in Medellin, Colombia — 123 is the emergency number in Colombia. The 123- woman line consists of supplementary emergency services to meet the demands of urgency in relation to cases of VAW. This service is implemented by the mayor of Medellin, in collaboration with the national police who is the institution in charge of managing the 123 line.
  When the police attends an emergency on VCM, the call is derived to the 123- woman line. There, a team consisting of a psychologist and a lawyer serves women in crisis, as emergency services provided by the police are developed in parallel. The team verifies that the rights of women are respected and that women are oriented to the relevant services. The 123- woman line operates from 7:00 am to 7:00 pm, Monday through Friday.
  Groups: 123 women line

SUMMARY:
The purpose of this study is to determine whether the 123 women emergency phone line of Medellin (Colombia) leads to a reduction in the violence suffered by women, as well as in their psychological wellbeing and attitudes towards violence.

DETAILED DESCRIPTION:
The purpose of this study is to determine whether the 123 women emergency phone line of Medellin (Colombia) leads to a reduction in the violence suffered by women, as well as in their psychological wellbeing and attitudes towards violence.

There is excess demand for the 123 women emergency phone line of Medellin. While on average 10 cases are reported (excluding referrals at night by the police, between 7pm and 7:00 a.m.), the average daily capacity of operation is 6 cases. So, is not possible for the 123 women team to track all women who call in 24 hours. Women who cannot receive the services of the 123 women team only get the emergency support of the police and do not receive additional aid (while it is verified that the rights of women are respected and they are guided to relevant services). The excess of demand over the capacity of the team of the 123 women line represents a natural experiment.

Women will be recruited from those who are attended by the 123 emergency women phone line immediately as well as from those who were only attended by emergency support of the police and may have received later the support of the 123 women line (control group). In a first instance, women will be called to verify their address. A face to face survey will be conducted by mid-2015.

ELIGIBILITY:
Inclusion Criteria:

* Women that call the 123 emergency line

Exclusion Criteria:

-

Ages: 18 Years to 65 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Women that call the 123 emergency line in Medellín, Colombia
Sampling Method: Probability Sample
Enrollment: 765 (Actual)
Dates: Start 2014-06; Primary Completion 2015-09 (Actual); Study Completion 2016-06 (Actual)

PRIMARY OUTCOMES:
Occurrence of violence | 3 months
  The outcome will be measure through a survey to women who called the 123 emergency line, some had besides the support of the police, immediate services from the 123 women line to have special services from a psychologist and a lawyer

SECONDARY OUTCOMES:
Knowledge, attitudes and practices (KAP) on violence and care pathways | Average of 6 months after calling the 123 emergency line
  The outcome will be measure through a survey to women who called the 123 emergency line, some had besides the support of the police, immediate services from the 123 women line to have special services from a psychologist and a lawyer
Psychological well-being (self-acceptance, positive relationships, autonomy, environmental mastery, personal growth, purpose in life) | Average of 6 months after calling the 123 emergency line
  The outcome will be measure through a survey to women who called the 123 emergency line, some had besides the support of the police, immediate services from the 123 women line to have special services from a psychologist and a lawyer
Formal complaints | 3 months
  The outcome will be measure through a survey to women who called the 123 emergency line, some had besides the support of the police, immediate services from the 123 women line to have special services from a psychologist and a lawyer

CONTACTS AND LOCATIONS:
Locations (1):
- Econometria Consultores, Bogotá, Colombia